CLINICAL TRIAL: NCT05497778
Title: A Phase 1b Study of Gemcitabine and Nab-paclitaxel in Combination With IM156 in Patients With Advanced Pancreatic Cancer.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0130; NCI-2022-06636 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Phase followed by a Dose Expansion Phase (Experimental): In the Dose Escalation Phase of the study, we will identify the RPD2 of IM156. Subsequently, we will evaluate IM156 at the RP2D (established in the Dose Expansion Phase) and gemcitabine + nab-paclitaxel in the Dose Expansion Phase.
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: IM156

INTERVENTIONS:
Drug: Gemcitabine — Given by IV (vein)
  Other Names: Gemcitabine Hydrochloride; GemzarÂ®
Drug: Nab paclitaxel — Given by IV (vein)
  Other Names: Paclitaxel (protein-bound); Abraxane, ABI-007
Drug: IM156 — Given by PO

SUMMARY:
To learn if adding a new medication, IM156, to treatment with gemcitabine and nab-paclitaxel is safe and tolerable. The ability of this combination to improve the success of this treatment for these patients will also be studied.

DETAILED DESCRIPTION:
Primary Safety Objective:

To evaluate the safety and tolerability of IM156 with Gem+NP in patients with metastatic PDAC

Exploratory Efficacy Objective:

To evaluate the efficacy of IM156 with Gem+NP in patients with metastatic PDAC

Exploratory Biomarker Objective:

To identify biomarkers that are predictive of response to IM156 (i.e., predictive biomarkers), are associated with progression to a more severe disease state (i.e., prognostic biomarkers), are associated with resistance to IM156, are associated with susceptibility to developing adverse events, can provide evidence of study treatment activity, or can increase the knowledge and understanding of disease biology.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfill all the following criteria:

* Ability to understand and the willingness to sign a written informed consent form (ICF).
* Male or female participants ≥ 18 years of age at the time of screening. Because no dosing or adverse event data are currently available on the use of IM156 in combination with Gem + NP in patients <18 years of age, children are excluded from this study.
* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma.
* Must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria [13], defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. The measurable lesion must be outside of a radiation field if the participant received prior radiation.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (see Appendix 1).
* Naïve to any prior treatment for metastatic disease, including chemotherapy, biological therapy, or targeted therapy.

  * Prior adjuvant therapy (including chemotherapy and/or radiotherapy) for pancreatic adenocarcinoma is permitted if neoadjuvant or adjuvant therapy was completed at least 6 months prior to study enrollment. Prior adjuvant therapy may include Gem or NP.
  * Participants initially diagnosed with localized pancreatic cancer who have undergone chemotherapy then resection and had no evidence of disease are eligible if relapse of metastatic disease has occurred and if the last dose of chemotherapy was received more than 6 months before study entry.
* Prior radiation therapy must have been completed at least 14 days before investigational product administration.
* Prior surgery that required general anesthesia or other major surgery as defined by the investigator must be completed at least 4 weeks before investigational product administration.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable viral load
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study (hormonal or barrier method of birth control; abstinence), for the duration of study participation, and 90 days after completion of IM156 administration.
* The effects of IM156 on the developing human fetus are unknown. For this reason, all women of child-bearing potential (refer to MDA Policy CLN 1114), which includes all female patients younger than 55 years, must meet one of the following inclusion criteria:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months)
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (follicle stimulating hormone and estradiol in menopausal range, who have received whole pelvic radiation therapy)
  * History of bilateral tubal ligation or another surgical sterilization procedure.)
  * Use of approved methods of birth control before the study, for the duration of study participation, 90 days after completion of IM156 administration, and for at least 6 months after the final dose of NP. Approved methods are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), tubal ligation or hysterectomy, patient/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. For all women of childbearing potential who do not meet one of the four criteria above, a negative serum pregnancy test will be required within 2 weeks prior to dosing.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL (in absence of growth factor support)
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥ 9.0 g/dl
  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN without hepatic metastasis and ≤ 5 x ULN with hepatic metastasis
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN without hepatic metastasis and ≤ 5 x ULN with hepatic metastasis
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Creatine clearance >50 as calculated by the Cockcroft Gault Formula
* Patients with new brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy. Patients who have undergone CNS directed treatment can be enrolled provided they show evidence of stable lesions (and no new lesions) with no evidence of tumor progression for at least 4 weeks after CNS-directed treatment. Patients do not require a baseline imaging, unless clinically indicated.

Exclusion Criteria:

* Patients with a current evidence of diabetes mellitus who are currently being treated with another biguanide (e.g., metformin)
* Patients who are currently being treated with the following medications, which are sensitive CYP2D6 substrates per FDA.gov (Drug Development and Interactions; Table of Substrates, Inhibitors, and Inducers): atomoxetine, desipramine, dextromethorphan , eliglustat(e), nebivolol, nortriptyline, perphenazine, tolterodine, R-venlafaxine
* Patients with a history of serious gastrointestinal bleeding within 6 weeks prior to screening or patients with any disease possibly affecting the absorption of oral agents (malabsorption syndrome, hemorrhagic gastric ulcer, etc.)
* Patients with suspected serious infectious diseases, intestinal paralysis, bowel obstruction, interstitial pneumonia, or pulmonary fibrosis.
* Patients with a history of alcohol or drug abuse within 12 weeks prior to screening
* The effects of IM156 on the developing human fetus are unknown. For this reason, women who are pregnant or breastfeeding are excluding from this study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patients with uncontrolled underlying medical conditions (e.g., interstitial lung disease, active infections requiring antibiotics, recent hospitalization with unresolved symptoms, symptomatic congestive heart failure [New York Heart Association class III or IV], unstable angina, uncontrolled hypertension, cardiac arrhythmia, interstitial lung disease, active coagulopathy).
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* History of myocardial infarction within 6 months or history of arterial thromboembolic event within 3 months of the first dose of investigational agent.
* Any active autoimmune disease.
* Any concurrent investigational anticancer therapy.
* Any concurrent immunosuppressive medications, including chronic systemic corticosteroids at greater than physiologic doses (a dose of 10 mg/day oral prednisone or equivalent) 14 days before the first dose (except for participants who require hormone replacement therapy such as hydrocortisone). A temporary course (≤ 3 days) of corticosteroids (i.e., contrast allergy, chronic obstructive pulmonary disease) may be permitted, depending on the duration and dose, after discussion and agreement with the PI.
* Any concurrent chemotherapy, radiotherapy (except palliative radiotherapy), immunotherapy, biologic, or hormonal treatment. Concurrent use of hormones for noncancer-related conditions is permitted.
* Patients who have not recovered from adverse events due to prior anticancer therapy (i.e., have residual toxicities > Grade 1) except for alopecia.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IM156, Gem or NP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 | through study completion and or average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Pant, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org